CLINICAL TRIAL: NCT00414596
Title: Pilot Study to Evaluate The Effectiveness And Safety Of Axiom Worldwide Drx9000™ Spinal Decompression System For Treatment of Low Back Pain
Brief Title: Pilot Study to Evaluate The Effectiveness And Safety Of Axiom Worldwide Drx9000™ Spinal Decompression System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NEMA Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-AXW01
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DRX Group (Experimental): Patients using the device DRX9000™.
  Interventions: Device: DRX9000™

INTERVENTIONS:
Device: DRX9000™ — Device is designed to apply spinal decompressive forces.

SUMMARY:
This pilot study will evaluate the effectiveness and safety of the Axiom Worldwide DRX9000 for active treatment of chronic low back pain.

DETAILED DESCRIPTION:
Currently, there are no prospective safety and/or outcomes studies utilizing the DRX9000™ in the peer-reviewed medical literature. There are published trials utilizing similar machines which provided evidence in support of the FDA granted indications for use spinal decompression and of the DRX9000™. Axiom Worldwide has determined it will be of benefit to the continuing medical care of patients and a furthering of the scientific knowledge of the treatment of LBP to complete such a prospective evaluation using a standardized treatment protocol. This study will therefore attempt to establish and validate the safety and efficacy of this computerized spinal decompression system in the treatment of LBP and sciatica.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, greater than 18 years of age
* Able to understand possible risks and benefits and provide written informed consent (ICF) to the IRB approved clinical multimodal protocol
* LBP with an intensity level of greater than 4 on an eleven point numerical pain rating scale (VRS) of 0-10 (with 0 - no pain and 10 - worst possible pain)
* Completed the necessary diagnostic and medical history evaluations as described in the protocol to confirm the patient's diagnosis and eligibility for the study and DRX9000 treatment protocol.
* Willing and able to complete a six week 20 session of DRX9000 outpatient treatments and a minimum of 6 months follow-up

Exclusion Criteria:

* Pregnancy
* Evidence of neurological motor deficits on clinical examination
* Evidence of spinal cord compression, metastatic cancer, tumor, hematoma, infection or compression fracture
* Evidence of severe central stenosis with neurological deficits or nerve root entrapment
* Litigation for health-related claim (in process or pending), Worker's Compensation, or Personal Injury
* Previous spine fusion surgery, insertion of hardware or artificial disc
* Hemiplegia or paraplegia
* History of severe cardiovascular or metabolic disease, or abdominal aortic aneurysm
* Unwillingness to postpone other types of therapy for LBP during the 6 week treatment sessions
* Known alcohol abuse or drug abuse
* Height less than 4 feet 10 inches (147 cm) or greater than 6 feet 8 inches (203 cm)
* Body weight greater than 300 pounds (136 kg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Leslie, MD, Principal Investigator — Mayo Clinic; Charlotte Richmond, PhD, Study Director — NEMA Research, Inc.; Joseph V Pergolizzi, MD, Study Chair — Naples Anesthesia and Pain Associates
Locations (3):
- United States (3):
  - Vibrance Medical Group, Beverly Hills, California
  - Naples Anesthesia and Pain Associates, Naples, Florida
  - Active Health and Wellness Center, Tampa, Florida

REFERENCES:
- See also: click here for more information about the DRX9000 — http://www.axiomworldwide.com
- See also: Nema Research website — http://www.nema.net

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DRX Group
Started | 20 (December 2006)
Completed | 18 (April 2007)
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | DRX Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Post-treatment Numerical Pain Intensity Rating Scale (VRS), Which is a Scale From 0-10 (0=no Pain, 10= Worst Pain)
Description: The numerical results of the post-treatment verbal numerical pain intensity rating scale (VRS) following completion of a standard six week series of 20 DRX9000 treatments.
Time Frame: Six weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DRX Group
Number analyzed (Participants) | 18
units on a scale | 0 [0 to 7]
Statistical Analysis 1: Comparison: DRX Group; Hypothesis: Patients with chronic low back pain who undergo spinal decompression with a standardized 6-week regimen consisting of 20 treatments with the spinal decompression system would experience >50% reduction in their verbal score of pain intensity. Power Analysis: Mean pain scores at time of enrollment were assumed to equal 6 with potential reduction in pain of 50%. To obtain 80% power at an alpha level of 0.05, sample size was estimated as 20 patients; Test type: Superiority or Other; p = .0001, Mixed Models Analysis; The primary pain end-point was assessed by a mixed effect model with time (visit) and as fixed effects and subject as random effect

2. Secondary Outcome: Recurrence for Significant (VRS Greater Than or Equal to 4) LBP Following Completion of 6 Weeks of DRX9000 Treatment.
Description: The number of Subjects reporting VRS greater than or equal to 4 for LBP following completion of 6 weeks of DRX9000 treatment will be recorded.
Time Frame: Six weeks
Measure: Number; unit: participants
Arm/Group | DRX Group
Number analyzed (Participants) | 18
participants | 1

3. Secondary Outcome: Change in Functional Capacity From Baseline to Six Weeks (The Revised Oswestry Pain Questionaire)
Description: Subject functional capacity following 6 weeks of DRX9000 treatment will be measured as a numerical score by the Revised Oswestry Pain Questionaire (scale 0-50, 0=pain without effects). Functional capacity was assessed at Baseline, 3 Weeks and 6 Weeks.
Time Frame: Six weeks
Measure: Median (Inter-Quartile Range); unit: Change in units of scale
Arm/Group | DRX Group
Number analyzed (Participants) | 18
Change in units of scale
  Baseline | 26 [7 to 34]
  Week 3 | 14 [0 to 26]
  Week 6 | 3 [0 to 26]

4. Secondary Outcome: Patient's Satisfaction With Treatment Procedures Following 6 Weeks of DRX9000 Treatment.
Description: Patient's satisfaction with treatment procedures following 6 weeks of DRX9000 treatment was measured on a scale from 0-10 (0= very unsatisfied, 10=very satisfied).
Time Frame: Six weeks
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | DRX Group
Number analyzed (Participants) | 18
units on a scale | 8.1 [0 to 10]

5. Secondary Outcome: Number of Adverse Events Following 6 Weeks of DRX9000 Treatment.
Description: Total number of adverse events reported following 6 weeks of DRX9000 treatment.
Time Frame: Six weeks
Population: All subjects enrolled were included in the analysis. No adverse events related to study device were reported.
Measure: Number; unit: Number of Adverse Events
Arm/Group | DRX Group
Number analyzed (Participants) | 20
Number of Adverse Events | 10

6. Secondary Outcome: Number of Patients Who Withdraw From Study.
Description: Total number of patients who withdrew during the 6 weeks of treatment.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | DRX Group
Number analyzed (Participants) | 20
participants | 2

ADVERSE EVENTS:
Arm/Group | DRX Group
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 8/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRX Group (N=20)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Head Colds (General disorders) | 2 (2)
Sinus Headaches (General disorders) | 2 (2)
Sinus Infection (Infections and infestations) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No